CLINICAL TRIAL: NCT00113113
Title: Phase I Study of Rubitecan (RFS 2000) in the Treatment of Cancer Patients With Organ Dysfunction
Brief Title: Study of Rubitecan in Cancer Patients With Renal or Hepatic Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFS 2000-40; SGI-RUB-040; RFS 2000-040
Record Dates: First submitted 2005-06-03; First posted 2005-06-06 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Tumors
Keywords: rubitecan; Orathecin; 9-nitrocamptothecin; solid tumors; organ dysfunction; renal dysfunction; hepatic dysfunction; RFS 2000
MeSH Terms: conditions — Neoplasms; Renal Insufficiency; Liver Diseases | interventions — rubitecan

INTERVENTIONS:
Drug: Rubitecan

SUMMARY:
Cancer patients with liver or renal dysfunction will be treated with rubitecan capsules to define the maximum tolerated dose and the dose-limiting toxicity in this patient population, and to perform pharmacokinetic studies of rubitecan in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years of age.
* The patient has histologically or cytologically proven malignancy recurrent or refractory to standard treatment or for which there is no standard therapy.
* The patient has measurable disease.
* The patient has sufficiently recovered from the acute toxic effects of previous chemotherapy, radiotherapy (no less than 3 weeks prior to randomization), and/or immunotherapy.
* The patient's estimated life expectancy is at least 8 weeks.
* The patient has a National Cancer Institute Common Toxicity Criteria (NCI CTC) Performance Status between 0 and 2.
* The patient has adequate bone marrow function.
* The patient must not have active central nervous system (CNS) metastases.

Exclusion Criteria:

* The patient has any serious, uncontrolled intercurrent illness or infection.
* The patient is receiving anti-retroviral therapy (HAART) for HIV infection.
* The patient is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2001-08

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - The Center for Cancer Care and Research, St Louis, Missouri